CLINICAL TRIAL: NCT02457546
Title: A Single-Blinded, Randomized, Controlled Study to Evaluate the Safety and Effectiveness of EVICEL® Fibrin Sealant (Human) Compared to a Hydrogel Sealant as an Adjunct to Sutured Dural Repair
Brief Title: The EVICEL® Neurosurgery Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIOS-14-002; 2014-003954-15 (EudraCT Number)
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: Fibrin sealant; CSF leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak; Cerebrospinal Fluid Otorrhea | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVICEL Fibrin Sealant (Experimental): EVICEL is a human plasma-derived fibrin sealant composed of two components - thrombin and fibrinogen
  Interventions: Biological: EVICEL Fibrin Sealant
- Hydrogel sealant (Active Comparator): The sealant is composed of two solutions, a polyethylene glycol (PEG) ester solution and a trilysine amine solution
  Interventions: Device: Hydrogel sealant

INTERVENTIONS:
Biological: EVICEL Fibrin Sealant
  Other Names: fibrin sealant
  Arms: EVICEL Fibrin Sealant
Device: Hydrogel sealant
  Arms: Hydrogel sealant

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of EVICEL® Fibrin Sealant (Human) for use as an adjunct to sutured dural repair in cranial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age undergoing craniotomy/craniectomy for pathological processes in the supratentorial region or posterior fossa
* Subjects or legally authorized representatives must be willing to participate in the study and provide written informed consent.
* Surgical wound classification Class I
* The cuff of native dura along the craniotomy edge on each side is adequate, based on surgeon's judgment, to facilitate suturing and to allow for sufficient surface area for adherence of the investigational product
* Presence of intra-operative cerebrospinal fluid (CSF) leakage following primary dural closure or after Valsalva maneuver

Exclusion Criteria:

* Subjects with a dural lesion from a recent surgery that still has the potential for CSF leakage.
* Chemotherapy within 30-days prior to enrollment or scheduled within 7-days following surgery
* Radiation therapy to the head within 30-days prior to enrollment or scheduled within 7-days following surgery
* A previous craniotomy/craniectomy within 6 months prior to the study surgery.
* Known hypersensitivity to the components of the investigational product.
* Subjects with a known allergy to FD&C Blue #1 dye
* Subjects with an infection present at the surgical site
* Subjects with an infection indicated by any one of the following: clinical diagnosis of infection, fever, positive urine culture, positive blood culture, positive chest X-ray.
* Female subjects of childbearing potential with a positive pregnancy test or intent to become pregnant during the clinical study period.
* Female subjects who are nursing.
* Exposure to another investigational drug or device clinical trial within 30 days prior to enrollment or anticipated in the 60 day follow-up period.
* Subjects with severely altered renal or hepatic function, with a compromised immune system or autoimmune disease who can NOT receive hydrogel sealant.
* Subjects with penetratring traumatic injuries to the head with damage to the dura
* Dural injury during craniotomy/craniectomy that cannot be eliminated by widening the craniotomy/craniectomy to recreate the native dural cuff.
* Patient has a gap between durotomy edges of greater than 2mm after primary dural closure.
* Approaches that would not allow sutured dural closure such as trans-sphenoidal or trans-labirinthine-/petrosal/-mastoid. Superficial penetration of mastoid air cells are allowed.
* Use of implants made of synthetic materials coming into direct contact with dura
* Use of other fibrin sealants or PEG-based sealants on the dural closure. Approved fibrin sealants may be used for hemostasis if not in contact with the dura.
* Hydrocephalus, except occlusive hydrocephalus caused by posterior fossa pathology or incompletely open cerebrospinal fluid pathways, to be treated during surgical procedure.
* Placement of Gliadel Wafers
* Intersecting durotomy scars in the surgical path from a previous operation that cannot be completely removed by the planned dural resection.
* Two or more separate cranial dural defects, including defects from ventricular cannulation and ventriculo-peritoneal shunting.
* Subjects with any other intra-operative findings identified by the surgeon that may preclude the conduct of the study procedure.
* Confined bony structures where nerves are present where neural compression may result due to swelling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kocharian, MD, PhD, Study Director — Ethicon, Inc.
Locations (26):
- United States (13):
  - Clinical Investigation Site #27, Los Angeles, California
  - Clinical Investigation Site #17, Sacramento, California
  - Clinical Investigation Site #18, Jacksonville, Florida
  - Clinical Investigation Site #19, Tampa, Florida
  - Clinical Investigation Site #22, Indianapolis, Indiana
  - Clinical Investigation Site #10, New Orleans, Louisiana
  - Clinical Investigation Site #15, Baltimore, Maryland
  - Clinical Investigation Site #11, Boston, Massachusetts
  - Clinical Investigation Site #24, Ann Arbor, Michigan
  - Clinical Investigation Site #20, New Brunswick, New Jersey
  - Clinical Investigation Site #12, New York, New York
  - Clinical Investigation Site #14, Cincinnati, Ohio
  - Clinical Investigation Site #21, Philadelphia, Pennsylvania
- Australia (4):
  - Clinical Investigation Site #51, Sydney, New South Wales
  - Clinical Investigation Site #54, Adelaide, South Australia
  - Clinical Investigation Site #50, Melbourne, Victoria
  - Clinical Investigation Site #52, Richmond, Victoria
- Belgium (2):
  - Clinical Investigation Site #40, Genk
  - Clinical Investigation Site #41, Leuven
- Clinical Investigation Site #25, Montreal, Quebec, Canada
- Clinical Investigation Site #53, Auckland, New Zealand
- United Kingdom (5):
  - Clinical Investigation Site #35, London, England
  - Clinical Investigation Site #32, Middlesbrough, England
  - Clinical Investigation Site #35, Nottingham, England
  - Clinical Investigation Site #30, Oxford, England
  - Clinical Investigation Site #31, Salford, England

REFERENCES:
- [Background] Green AL, Arnaud A, Batiller J, Eljamel S, Gauld J, Jones P, Martin D, Mehdorn M, Ohman J, Weyns F. A multicentre, prospective, randomized, controlled study to evaluate the use of a fibrin sealant as an adjunct to sutured dural repair. Br J Neurosurg. 2015 Feb;29(1):11-17. doi: 10.3109/02688697.2014.948808. Epub 2014 Aug 12. PMID 25112563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from medical centers in North America, Europe, and Asia-Pacific. The first subject was randomized on July 7 2015 and the last subject completed the study October 12 2017
Groups:
- Evicel: EVICEL® is a human plasma-derived fibrin sealant. EVICEL® consists of two components: a concentrate of Human Fibrinogen (referred to as Biological Component 2; BAC2) and a solution of Human Thrombin, which incorporates calcium.
- DuraSeal: DuraSeal™ Dural Sealant System is a commercially available synthetic sealant intended for use as an adjunct to sutured dural repair during cranial surgery to provide watertight closure. The product is a synthetic absorbable sealant composed of a polyethylene glycol (PEG) ester solution and a rilysine amine solution.
Period: Overall Study
Arm/Group | Evicel | DuraSeal
Started | 114 | 120
Completed | 105 | 116
Not Completed | 9 | 4
Not completed — Other reasons | 4 | 1
Not completed — Refused to complete study/procedures | 1 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data was summarized for the intent to Treat (ITT) Set, which included all randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Evicel | DuraSeal | Total
Number analyzed (Participants) | 114 | 120 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (14.9) | 56.0 (15.0) | 54.7 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 55 | 61 | 116
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 102 | 101 | 203
  Black or African American | 9 | 9 | 18
  American Indian or Alaska Native | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Asian | 1 | 2 | 3
  Other | 1 | 4 | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (6.0) | 26.9 (5.0) | 27.2 (5.5)
BMI (Grouped) [Count of Participants; unit: Participants] — Description: Underweight: < 18.5 kg/m^2, normal weight: 18.5 - < 25kg kg/m^2, Overweigh: 25 - < 30 kg/m^2, Obese: 30 - < 40 kg/m^2, Morbidly obese: 40 kg/m^2 or more
  Participants
    Underweight | 1 | 1 | 2
    Normal | 37 | 46 | 83
    Overweight | 45 | 39 | 84
    Obese | 27 | 34 | 61
    Morbidly Obese | 4 | 0 | 4
Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 2 | 3 | 5
  Non-Hispanic | 112 | 117 | 229

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint Success Number of Successes (Subjects That Had no Inter-operative CSF Leak Following Valsalva Maneuver and no CSF Leak or Pseudomeningocele in the Surgical Area During the 30-day Follow-up Period)
Description: The primary endpoint was the proportion of subjects that had no inter-operative CSF leak following Valsalva maneuver and no CSF leak or pseudomeningocele in the surgical area during the 30-day follow-up period
Time Frame: Intraoperatively through 30-day follow-up
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Arm/Group | Evicel | DuraSeal
Number analyzed (Participants) | 102 | 106
Participants
  Posterior Fossa: number analyzed (Participants) | 27 | 29
  Posterior Fossa | 22 | 23
  Supratentorial: number analyzed (Participants) | 75 | 77
  Supratentorial | 73 | 69
  Total | 95 | 92
Statistical Analysis 1: Comparison: Evicel vs DuraSeal; Test type: Non-Inferiority — The statistical hypothesis for testing the treatment difference was presented as follows: H0: Δ ≤ -0.10 tested against the alternative hypothesis Ha: Δ > -0.10. where: * Δ is the difference between the success rates of Experimental (Evicel®) and Control (DuraSeal™) (Experimental minus Control) * -0.10 is the non-inferiority difference PC is the proportion of success in DuraSeal™ Control subjects and PE is the proportion of success in EVICEL® subjects; Difference in Success Rates = 6.3, 95% CI 2-sided [-1.8 to 14.4]

2. Other Pre Specified Outcome: Safety Endpoint: Intra-operative CSF Leakage Follow Final Valsalva
Description: Intra-operative CSF leakage follow final Valsalva
Time Frame: Intraoperatively, after final Valsalva maneuver
Population: No Valsalva maneuver performed in 2 participants in the Evicel Arm and 1 participant in the DuraSeal Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Evicel | DuraSeal
Number analyzed (Participants) | 112 | 119
Participants | 10 | 13

ADVERSE EVENTS:
Time Frame: From surgical procedure through the 60 day follow-up visit
Arm/Group | Evicel | DuraSeal
All-Cause Mortality (participants affected / at risk) | 3/114 | 2/120
Serious Adverse Events (participants affected / at risk) | 32/114 | 37/120
Other Adverse Events (participants affected / at risk) | 103/114 | 109/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evicel (N=114) | DuraSeal (N=120)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Brain empyema (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 3
Postoperative wound infection (Infections and infestations) | 2 | 5
Propionibacterium infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 2 | 9
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
White blood cell count increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 5
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Subdural hygroma (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Subgaleal haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evicel (N=114) | DuraSeal (N=120)
Tachycardia (Cardiac disorders) | 5 | 6
Constipation (Gastrointestinal disorders) | 32 | 29
Nausea (Gastrointestinal disorders) | 32 | 29
Vomiting (Gastrointestinal disorders) | 20 | 14
Chest pain (General disorders) | 5 | 6
Fatigue (General disorders) | 4 | 6
Pyrexia (General disorders) | 3 | 10
Pneumonia (Infections and infestations) | 5 | 6
Postoperative wound infection (Infections and infestations) | 4 | 6
Incision site pain (Injury, poisoning and procedural complications) | 11 | 12
Procedural pain (Injury, poisoning and procedural complications) | 19 | 19
Pseudomeningocele (Injury, poisoning and procedural complications) | 2 | 9
Wound secretion (Injury, poisoning and procedural complications) | 6 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Convulsion (Nervous system disorders) | 3 | 9
Dizziness (Nervous system disorders) | 5 | 10
Headache (Nervous system disorders) | 37 | 54
Hemiparesis (Nervous system disorders) | 7 | 3
Confusional state (Psychiatric disorders) | 0 | 7
Hypertension (Vascular disorders) | 12 | 12
Hypotension (Vascular disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/46/NCT02457546/SAP_000.pdf
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02457546/Prot_001.pdf